CLINICAL TRIAL: NCT07264998
Title: Gut Microbiota Changes in Breast Cancer Patients Treated With Abemaciclib and Correlation With Drug-Induced Diarrhea: An Observational Cohort Study
Brief Title: Observational Study of Gut Microbiota in Abemaciclib-Treated Patients With and Without Diarrhea
Status: Not yet recruiting | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xinhong Wu, PhD, vice-president, Hubei Cancer Hospital
Other Study IDs: LLHBCH2025YN-088
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasms; Hormone Receptor-Positive Breast Cancer; Abemaciclib; Abemaciclib-related Diarrhea; Drug-induced Diarrhea; Gastrointestinal Microbiome (Focus); Microbiome
Keywords: Abemaciclib; Hormone receptor-positive breast cancer; Drug-induced diarrhea; Microbiome; Gastrointestinal microbiome; Microbiome biomarkers; Abemaciclib-related diarrhea
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will retain the following types of biospecimens for future research:
  Fecal Samples: Approximately 5 grams of fresh stool will be collected from each participant using sterile containers. Samples will be stored at -80°C and may be used for DNA extraction, metagenomic sequencing, and other microbiome analyses.
  Blood Samples: Approximately 5 mL of peripheral blood will be collected via venipuncture. Serum will be separated, aliquoted, and stored at -80°C for potential future analyses, including metabolomic profiling, inflammatory cytokine measurement (e.g., IL-6, TNF-α, CRP), and other biomarker studies.
  All biospecimens will be de-identified and labeled with a unique study code to ensure participant confidentiality. Samples may be used to extract DNA and for other molecular analyses related to understanding the relationship between gut microbiota and drug-induced diarrhea.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Abema-Diarrhea: HR-positive breast cancer patients who develop diarrhea (Grade 1 or higher as per CTCAE v5.0 criteria) during treatment with Abemaciclib. This group will not receive any investigational intervention as part of the observational study. Fecal and blood samples will be collected for microbiome and biomarker analysis.
- Abema-NoDiarrhea: HR-positive breast cancer patients who do not develop diarrhea (Grade 0 as per CTCAE v5.0 criteria) during treatment with Abemaciclib. This group serves as the control cohort and will not receive any investigational intervention as part of the observational study. Fecal and blood samples will be collected for microbiome and biomarker analysis.

SUMMARY:
Why is this study being done? Many patients with a type of breast cancer (called HR-positive) take a medicine called Abemaciclib. While this medicine is effective, a very common side effect is diarrhea, which can be severe enough to disrupt treatment and reduce quality of life. The reason why some patients get diarrhea and others do not is not well understood. This study aims to investigate whether the natural bacteria living in the gut (known as the gut microbiome) play a role in this side effect. Researchers will compare the gut bacteria of patients who develop diarrhea with those who do not.

What will happen in the study? This is an observational study, which means that patients will receive their normal cancer treatment and will not be given any new or experimental drugs as part of this initial phase.

* Patients who are already being treated with Abemaciclib will be invited to join.
* They will be placed into one of two groups: those who experience diarrhea and those who do not.
* Participants will be asked to provide stool (feces) samples and may also provide optional blood samples at specific times during their treatment.
* Researchers will analyze these samples in the lab to study the types and functions of the gut bacteria.

Who can participate?

* Adult women (aged 18-75) diagnosed with HR-positive breast cancer.
* Currently receiving treatment with Abemaciclib for at least 2 weeks.
* Must be willing to provide informed consent and follow the study procedures.

What are the potential benefits? Participants will not receive any direct medical benefit from taking part in this study. However, the information learned may help researchers better understand why diarrhea occurs and, in the future, could lead to new ways to prevent or treat this side effect for other cancer patients.

How is privacy protected? All personal information and samples collected will be de-identified using a unique code. This means that the data used for analysis cannot be directly linked back to the participant's identity. All data is stored securely according to strict ethical guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years.
2. Diagnosed with hormone receptor-positive (HR⁺) breast cancer.
3. Currently receiving treatment with Abemaciclib (either as monotherapy or in combination with endocrine therapy) for a duration of at least 2 weeks.
4. Willing and able to provide written informed consent for participation in the study.

Exclusion Criteria:

1. History of major gastrointestinal diseases, such as inflammatory bowel disease, Crohn's disease, ulcerative colitis, or intestinal obstruction, or having undergone major gastrointestinal surgery.
2. Recent use (within 1 month) of antibiotics, probiotics, or traditional Chinese medicine that may alter gut function.
3. Pregnant or lactating women.
4. Unwilling to provide informed consent or considered by the investigator to be unsuitable for the study for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll a prospective cohort of female patients with hormone receptor-positive (HR⁺) breast cancer who are receiving treatment with Abemaciclib (as monotherapy or in combination) as part of their standard clinical care at Hubei Cancer Hospital. Participants will be prospectively assigned into two groups based on the presence or absence of drug-induced diarrhea, as defined by CTCAE v5.0 criteria: the Diarrhea Group and the Non-Diarrhea (Control) Group. The study involves the collection of clinical data, fecal samples, and optional blood samples for microbiome and biomarker analysis. No investigational intervention is administered in this phase of the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in gut microbiota beta diversity | Through study completion, an average of 6 months.
  Beta diversity of the gut microbiome (e.g., Weighted UniFrac distance) will be compared between the diarrhea group and the non-diarrhea group to assess overall microbial community structure differences.
Identification of specific bacterial species enriched in non-diarrhea group | Through study completion, an average of 6 months.
  Metagenomic sequencing data will be analyzed (e.g., using LEfSe) to identify bacterial species that are significantly enriched in the non-diarrhea group compared to the diarrhea group (LDA Score > 2, p-value < 0.05).

SECONDARY OUTCOMES:
Difference in gut microbiota alpha diversity | Through study completion, an average of 6 months.
  Alpha diversity indices (Shannon, Chao1) of the gut microbiome will be compared between the diarrhea group and the non-diarrhea group.
Difference in metagenomic functional pathways | Through study completion, an average of 6 months.
  Differential abundance analysis of functional pathways (e.g., KEGG Level 2/3) derived from metagenomic sequencing data between the two groups.
Differential metabolites in serum | Through study completion, an average of 6 months.
  Differences in serum metabolomic profiles between the diarrhea and non-diarrhea groups.
Difference in systemic inflammatory cytokine levels | Through study completion, an average of 6 months.
  Levels of inflammatory cytokines (e.g., IL-6, TNF-α, CRP) in serum will be compared between the two groups.

OTHER OUTCOMES:
Predictive potential of baseline gut microbiota | Through study completion, an average of 6 months.
  Exploratory analysis to assess the potential of baseline gut microbiota features for predicting the risk of developing Abemaciclib-induced diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) that underlie the results reported in this study will not be shared publicly. The decision is based on the following considerations: to protect patient privacy and confidentiality, as the data contain sensitive clinical and genomic information; the informed consent obtained from participants does not include provisions for public data sharing; and the samples and data are collected under a specific ethical approval that limits their use to this research protocol. Summary results and aggregated data will be made available through publication.